CLINICAL TRIAL: NCT06819397
Title: Effects of Post-Isometric Relaxation Technique Versus Cross Friction Soft Tissue Mobilization on Pain, Range of Motion, and Endurance in Leg Spin Bowlers With Rotator Cuff Strain
Brief Title: Effects of Post-Isometric Relaxation Technique Vs Soft Tissue Mobilization in Leg Spin Bowlers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0406
Record Dates: First submitted 2025-01-22; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Sports Physical Therapy
Keywords: cross friction soft tissue mobilization, spin bowlers

STUDY DESIGN:
Intervention Model Description: parallel assignment randomized clinical design
Who Masked: Participant
Masking Description: single (participant) the participants are blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- post isometric relaxation (Experimental): 17 participants will be in post isometric group, After telling the bowler to calm down, a fresh movement barrier will be activated. This will be done three times a week for four weeks, for a total of five sets of five repetitions.
  Interventions: Other: post isometric relaxation
- cross friction soft tissue mobilization (Experimental): 17 participants will be in soft tissue mobilization group, Patients in each group will receive12 treatment sessions, 3 days a week for 4 weeks.
  Interventions: Other: cross friction soft tissue mobilization

INTERVENTIONS:
Other: post isometric relaxation — the athlete will be given instructions to perform a 7-second isometric contraction in the direction of horizontal abduction at about 25% of peak effort, while the examiner will apply an opposing force at the distal humerus.
  Arms: post isometric relaxation
Other: cross friction soft tissue mobilization — by identifying the fascia restriction, patients in group B will be treated with the cross friction soft tissue mobilization approach, which comprised applying a low load and prolonged stretch through the knuckles or elbows to the constricted fascia. The therapist will then give the contralateral side of rotation resistance for ten seconds
  Arms: cross friction soft tissue mobilization

SUMMARY:
Effects of Post-Isometric Relaxation Technique versus Cross Friction Soft Tissue Mobilization in Leg Spin Bowlers with Rotator cuff strain

DETAILED DESCRIPTION:
The existing body of research on Pakistani Cyclists lacks comprehensive investigation into the role of sciatic nerve flossing and active release technique, creating a noticeable gap in understanding the impact of such techniques on the performance, improving flexibility, and overall physical well-being of these athletes. Given the unique physical demands of Cyclists and the potential benefits associated with lower limb muscle strength, a focused exploration in this area is crucial to inform training strategies, enhance athletic performance, and contribute to the holistic development of Pakistani cyclists. To determine the comparative impact of sciatic nerve flossing and active release technique on pain, flexibility, and functionality in the lower limbs of cyclists with sciatica.

ELIGIBILITY:
Inclusion Criteria:

* age 16-30 years
* Symptomatic male bowlers (leg spinners)
* Pain from at least 2 months
* Playing regularly from at least 1 year.
* Difference of ROM as compared to contralateral extremity.

Exclusion Criteria:

* Prior History of shoulder surgery
* Shoulder symptoms requiring medical treatment.
* Cricketers not involved in any other sports.

Ages: 16 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS): | 4weeks
  The patient's degree of pain is measured using the 11-point NPRS. The words "no pain" on the left and "worst imaginable pain" on the right serve as the scale's anchors. (34) Patients score how much pain they are in right now, as well as how much pain they have had in the past 24 hours.
Goniometer | 4weeks
  Studies have shown intra-rater reliability for goniometric measurements can vary but often falls within acceptable ranges. For instance, a study reported intra-rater reliability with an intra-class correlation coefficient (ICC) ranging from 0.80 to 0.95, indicating good to excellent reliability.
Standard test for push-up (STPU) for measuring endurance | 4weeks
  Standard push-up test (STPU)" starts from either a prone position or a straight arm support position. Arms are about shoulder-width apart, palms are flat on the ground, and fingers are pointing forward. Legs should be together, ankles flexed, and knees locked. The only parts of the body that touch the ground are the balls of the feet and the palms of the hands. Until the chin, nose, or chest reaches the ground, the body is lowered.

CONTACTS AND LOCATIONS:
Overall Officials: Saad Arif, DPT, Principal Investigator — Riphah International University
Locations (1):
- Jallo Cricket Academy, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pandey V, Jaap Willems W. Rotator cuff tear: A detailed update. Asia Pac J Sports Med Arthrosc Rehabil Technol. 2015 Feb 11;2(1):1-14. doi: 10.1016/j.asmart.2014.11.003. eCollection 2015 Jan. PMID 29264234
- [Background] Hermans J, Luime JJ, Meuffels DE, Reijman M, Simel DL, Bierma-Zeinstra SM. Does this patient with shoulder pain have rotator cuff disease?: The Rational Clinical Examination systematic review. JAMA. 2013 Aug 28;310(8):837-47. doi: 10.1001/jama.2013.276187. PMID 23982370
- [Background] Jain NB, Wilcox RB 3rd, Katz JN, Higgins LD. Clinical examination of the rotator cuff. PM R. 2013 Jan;5(1):45-56. doi: 10.1016/j.pmrj.2012.08.019. PMID 23332909
- [Background] Tawfik AM, El-Morsy A, Badran MA. Rotator cuff disorders: How to write a surgically relevant magnetic resonance imaging report? World J Radiol. 2014 Jun 28;6(6):274-83. doi: 10.4329/wjr.v6.i6.274. PMID 24976930
- [Background] Shaffer B, Huttman D. Rotator cuff tears in the throwing athlete. Sports Med Arthrosc Rev. 2014 Jun;22(2):101-9. doi: 10.1097/JSA.0000000000000022. PMID 24787724
- [Background] Avci O, Rohrle O. Determining a musculoskeletal system's pre-stretched state using continuum-mechanical forward modelling and joint range optimization. Biomech Model Mechanobiol. 2024 Jun;23(3):1031-1053. doi: 10.1007/s10237-024-01821-x. Epub 2024 Apr 15. PMID 38619712
- [Background] Coviello JP, Kakar RS, Reynolds TJ. SHORT-TERM EFFECTS OF INSTRUMENT-ASSISTED SOFT TISSUE MOBILIZATION ON PAIN FREE RANGE OF MOTION IN A WEIGHTLIFTER WITH SUBACROMIAL PAIN SYNDROME. Int J Sports Phys Ther. 2017 Feb;12(1):144-154. PMID 28217425
- [Background] Bailey LB, Shanley E, Hawkins R, Beattie PF, Fritz S, Kwartowitz D, Thigpen CA. Mechanisms of Shoulder Range of Motion Deficits in Asymptomatic Baseball Players. Am J Sports Med. 2015 Nov;43(11):2783-93. doi: 10.1177/0363546515602446. Epub 2015 Sep 24. PMID 26403207
- [Background] Kim J, Sung DJ, Lee J. Therapeutic effectiveness of instrument-assisted soft tissue mobilization for soft tissue injury: mechanisms and practical application. J Exerc Rehabil. 2017 Feb 28;13(1):12-22. doi: 10.12965/jer.1732824.412. eCollection 2017 Feb. PMID 28349028
- [Background] Cunningham G, Charbonnier C, Ladermann A, Chague S, Sonnabend DH. Shoulder Motion Analysis During Codman Pendulum Exercises. Arthrosc Sports Med Rehabil. 2020 Jun 26;2(4):e333-e339. doi: 10.1016/j.asmr.2020.04.013. eCollection 2020 Aug. PMID 32875297
- [Background] Bhosale P, Kolke Pt S. Effectiveness of instrument assisted soft tissue mobilization (IASTM) and muscle energy technique (MET) on post-operative elbow stiffness: a randomized clinical trial. J Man Manip Ther. 2023 Oct;31(5):340-348. doi: 10.1080/10669817.2022.2122372. Epub 2022 Sep 28. PMID 36171728
- [Background] Khan ZK, Ahmed SI, Baig AAM, Farooqui WA. Effect of post-isometric relaxation versus myofascial release therapy on pain, functional disability, rom and qol in the management of non-specific neck pain: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Jun 13;23(1):567. doi: 10.1186/s12891-022-05516-1. PMID 35698187
- [Background] Cheatham SW, Stull KR, Kolber MJ. Roller massage: is the numeric pain rating scale a reliable measurement and can it direct individuals with no experience to a specific roller density? J Can Chiropr Assoc. 2018 Dec;62(3):161-169. PMID 30662071
- [Background] Shamsi M, Mirzaei M, Khabiri SS. Universal goniometer and electro-goniometer intra-examiner reliability in measuring the knee range of motion during active knee extension test in patients with chronic low back pain with short hamstring muscle. BMC Sports Sci Med Rehabil. 2019 Mar 22;11:4. doi: 10.1186/s13102-019-0116-x. eCollection 2019. PMID 30949343
- [Background] van Rijn SF, Zwerus EL, Koenraadt KL, Jacobs WC, van den Bekerom MP, Eygendaal D. The reliability and validity of goniometric elbow measurements in adults: A systematic review of the literature. Shoulder Elbow. 2018 Oct;10(4):274-284. doi: 10.1177/1758573218774326. Epub 2018 Jun 3. PMID 30214494
- [Background] Kiatkulanusorn S, Luangpon N, Srijunto W, Watechagit S, Pitchayadejanant K, Kuharat S, Beg OA, Suato BP. Analysis of the concurrent validity and reliability of five common clinical goniometric devices. Sci Rep. 2023 Nov 27;13(1):20931. doi: 10.1038/s41598-023-48344-6. PMID 38017058
- [Background] Rodrigues da Silva Barros B, Dal'Ava Augusto D, de Medeiros Neto JF, Michener LA, Silva RS, Sousa CO. Isometric versus isotonic exercise in individuals with rotator cuff tendinopathy-Effects on shoulder pain, functioning, muscle strength, and electromyographic activity: A protocol for randomized clinical trial. PLoS One. 2023 Nov 13;18(11):e0293457. doi: 10.1371/journal.pone.0293457. eCollection 2023. PMID 37956135